CLINICAL TRIAL: NCT03773042
Title: A Phase IIa, Multi-center, Open-label, Non-randomized, Active-controlled, and Dose-escalation Clinical Study Evaluating Tolerability, Efficacy, and Safety of HSK3486 Injectable Emulsion for Sedation/Anesthesia in Patients Undergoing Diagnostic Colonoscopy
Brief Title: A Study Evaluating Tolerability, Efficacy, and Safety of HSK3486 Injectable Emulsion in Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sichuan Haisco Pharmaceutical Group Co., Ltd (Industry)
Responsible Party: Sponsor
Organization: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HSK3486-201
Record Dates: First submitted 2018-12-06; First posted 2018-12-12 (Actual); Last update posted 2018-12-13 (Actual); Status verified 2017-06

CONDITIONS: Colonoscopy
MeSH Terms: interventions — HSK3486; Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HSK3486 (Experimental): 0.1mg/kg, 0.2mg/kg, 0.3mg/kg, 0.4mg/kg, 0.5mg/kg
  Interventions: Drug: HSK3486
- Propofol (Active Comparator): 1.0mg/kg, 2.0mg/kg
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: HSK3486 — For induction and maintenance of sedation.
  Arms: HSK3486
Drug: Propofol — For induction and maintenance of sedation.
  Arms: Propofol

SUMMARY:
A double-blind, randomized, active controlled, multi-center, parallel group study comparing HSK3486 with Propofol, in patients undergoing a colonoscopy.

ELIGIBILITY:
Inclusion Criteria (those who meet all of the following are eligible)

1. Patients requiring diagnostic colonoscopy with an estimated examination time ≤ 30 min; males and females, ASA grade I-II, between 18 and 65 years old (inclusive);
2. Body mass index (BMI) ≥ 18 and ≤ 30 kg/m2
3. Respiratory rate between ≥ 10 and ≤ 24 breaths per minute; SpO2 when inhaling > 95%; SBP ≥ 90 mmHg; DBP ≥ 60 mmHg; heart rate between ≥ 50 and ≤ 100 beats per minute;
4. Subjects must understand the procedures and methods of this study, and be willing to provide informed consent and to complete the trial in strict accordance with clinical trial protocol.

Exclusion Criteria (those who meet any one of the following are ineligible):

1. Patients having contraindications to general anesthesia or previous history of anesthesia accidents;
2. Patients with a known sensitivity to propofol, opioids, naloxone, eggs, soy products or a medical condition such that these agents were contraindicated;
3. Patient received any of the following drugs or therapies prior to screening:

   1. Participated in other drug clinical trials within 3 month prior to screening;
   2. In receipt of propofol and/or opioid analgesics within 1 month prior to screening;
4. The patient has some history or evidence of increased risk of sedation or anesthesia, such as cardiovascular disease, respiratory disease, cerebrovascular disease, gastrodintestinal disease and other system disease prior to the screening and/or baseline period.
5. Patient whose laboratory parameters measured at screening/prior to enrollment reach the following criteria and verified through re-examinations:

   1. ANC ≤ 1.5 x 109/L;
   2. PLT ≤ 80 x 109/L;
   3. Hb ≤ 90 g/L (no blood transfusion within the last 14 days);
   4. AST and ALT ≥ 2.5 x ULN;
   5. TBIL ≥ 1.5 x ULN;
   6. Creatinine ≥ 1.5 x ULN.
6. History of alcohol abuse within 3 months prior to screening or with a positive result of alcohol saliva strip test (before dose);
7. History of medication abuse within 3 months prior to screening, or a positive urine medication test (during screening or before dose administration);
8. Women who are pregnant or breastfeeding; women of child-bearing potential or men who are unwilling to use contraception during the trial; Patients who are planning pregnancy within 1 month after the completion of the trial (including male patients);
9. Potential difficult airway or difficult tracheal intubation, as determined by the investigator, and/or history of intubation failure;
10. Patients determined by the investigator to be unsuitable for participating in this trial for any reason.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Rate of successful colonoscopies. | From the first dose of the study drug to removal of colonoscope on day 1

SECONDARY OUTCOMES:
Insertion time | From the first dose of study drug until insertion of colonoscope on day 1
The success rate of the colonoscopy procedure | From the first dose of the study drug to removal of colonoscope on day 1
  The number of patients who successfully completed the colonoscopy procedure accounted for the proportion of all patients in the dose group
Time to fully alert | From the removal of colonoscopy procedure, until the first of three consecutive MOAA/S scores of 5 on day 1
Time to discharge | From the removal of colonoscopy procedure, until the first of three consecutive MOAA/S scores of 9 on day 1
Application of study drug and alternative medication | During the colonoscopy procedure on day 1
  Total dosages of study drug and alternative medication
Mini-Mental State Examinations (MMSE) | During the screening and the colonoscopy procedure on day 1

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No